CLINICAL TRIAL: NCT05341570
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BPI-21668 in Advanced Solid Tumor Patients
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BPI-21668
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTP-661511
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Oral tablets taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 28 days in duration with BPI-21668 administered, once daily (QD).
  Interventions: Drug: BPI-21668
- Dose Expansion (Experimental): Oral tablets administered at MTD/RP2D. Each treatment cycle will be 28 days in duration with BPI-21668 administered, once daily (QD).
  Interventions: Drug: BPI-21668

INTERVENTIONS:
Drug: BPI-21668 — Subjects will receive BPI-21668 until disease progression

SUMMARY:
This study is an open-label, single arm, dose escalation and dose expansion phase 1 study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of BPI-21668 in solid tumor patients. In dose escalation phase, biomarker status is not required, but in dose expansion phase patients are required to harbor PIK3CA mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤70 years, male and female patients;
2. Life expectancy ≥ 12 weeks;
3. ECOG performance score 0-1;
4. Locally advanced or relapsed/metastatic solid tumor patients, who had disease progression after standard therapy, intolerable to standard therapy or for whom no standard therapy exists, PIK3CA mutation status is required for dose expansion phase;
5. Evaluable lesion required for dose escalation phase and measurable lesion as per RECIST 1.1 required for dose expansion phase;
6. Adequate organ function;
7. Signed informed consent.

Exclusion Criteria:

1. Prior use of PI3K、mTOR or AKT inhibitor;
2. Prior other malignant tumor;
3. Unstable, symptomatic primary CNS tumors/metastasis or leptomeningeal metastases ;
4. Type I or type II diabetes;
5. Inadequate wash-out of prior anti-cancer therapies;
6. Cardiac disorders;
7. Instable systemic diseases;
8. Acute or chronic pancreatitis;
9. Pregnancy or lactation;
10. Other protocol specified criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The adverse events (AEs) | Through the Phase I, approximately 24 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events (AEs).
Determine the Maximum Tolerated Dose (MTD) | Through the Phase I, approximately 24 months
  The MTD will be based on DLT.
Determine the recommended Phase II dose (RP2D) | Through the Phase I, approximately 24 months
  The RP2D will be based on DLT.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of BPI-21668 | Through the Phase I, approximately 24 months
  Based on blood plasma concentration
Determination of anti-tumor activity of BPI-21668 | Through the Phase I, approximately 24 months
  Efficacy assessments (tumor evaluation) will be performed per RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No